CLINICAL TRIAL: NCT01931631
Title: A Practice-Based, Nutrition Intervention in Type 2 Diabetes
Brief Title: Plant-Based Dietary Intervention in Type 2 Diabetes-2
Acronym: WCCR-DIAB2
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was never initiated.
Sponsor: Physicians Committee for Responsible Medicine (Other)
Collaborators: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: PCRM GWU DM Study-2
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Diet, Vegetarian; Diet, Fat-Restricted; Glycemic Index
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet, Fat-Restricted; Diet, Vegan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Low-fat, low-Glycemic Index, vegan diet (Experimental): Low-fat, low-Glycemic Index, vegan diet
  Interventions: Behavioral: Low-fat, low-Glycemic Index, vegan diet
- ADA diet (Active Comparator): American Diabetes Association diet
  Interventions: Behavioral: ADA diet

INTERVENTIONS:
Behavioral: Low-fat, low-Glycemic Index, vegan diet — Low-fat, low-Glycemic Index, vegan diet
  Arms: Low-fat, low-Glycemic Index, vegan diet
Behavioral: ADA diet — Diet in accordance with the American Diabetes Association
  Arms: ADA diet

SUMMARY:
The purpose of the study is to assess whether, in individuals with type 2 diabetes, a low-fat, vegan diet improves blood glucose control more effectively than a control diet based on current American Diabetes Association (ADA) guidelines. The principal measure is hemoglobin A1c. Cardiovascular risk factors and dietary acceptability are also assessed. The study duration is 20 weeks with a one-year follow-up.

DETAILED DESCRIPTION:
Preliminary evidence suggests that low-fat, vegetarian regimens similar to those used to reverse coronary artery blockages may have a significant beneficial effect on type 2 diabetes, as demonstrated by reductions in fasting serum glucose concentrations and medication use. The investigators therefore randomly assigned 99 individuals with type 2 diabetes to either a low-fat, vegan diet or a diet based on current American Diabetes Association guidelines for 22 weeks with a one-year follow-up period. The principal dependent measure is hemoglobin A1c. Cardiovascular risk factors are also being tracked, as is dietary acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus

Exclusion Criteria:

- hemoglobin A1c values <6.5% or >10.5% use of insulin for > 5 years tobacco use within the preceding 6 months consumption of more than 2 alcoholic beverages per day current drug abuse pregnancy unstable medical status current use of a low-fat, vegetarian diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c | 20 weeks

SECONDARY OUTCOMES:
Body Weight | 20 Weeks
Blood Pressure | 20 Weeks
Glucose | 20 Weeks
Comprehensive Metabolic Panel | 20 Weeks & one-year follow up
Serum cholesterol and triacylglycerol concentrations | 20 Weeks
Urinary albumin and creatinine | 20 Weeks
Genotyping for Taq1 A and Taq1 B polymorphisms, and APOE (Apolipoprotein E) | 20 Weeks
Waist and hip circumference | 20 Weeks
Dietary Acceptability | 20 Weeks
3-day dietary records | 20 Weeks
International Physical Activity Questionnaire | 20 Weeks
Food Acceptability Questionnaire | 20 Weeks
Eating Inventory | 20 Weeks
CESD-R (Center for Epidemiologic Studies Depression Scale: Review and revision) | 20 Weeks
Beck Depression Inventory II (BDI-II) | 20 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Cohen, MD, Principal Investigator — George Washington University
Locations (1):
- Physicians Committee for Responsible Medicine, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
No data was collected because the study was never initiated.

REFERENCES:
- [Background] Ornish D, Scherwitz LW, Billings JH, Brown SE, Gould KL, Merritt TA, Sparler S, Armstrong WT, Ports TA, Kirkeeide RL, Hogeboom C, Brand RJ. Intensive lifestyle changes for reversal of coronary heart disease. JAMA. 1998 Dec 16;280(23):2001-7. doi: 10.1001/jama.280.23.2001. PMID 9863851
- [Background] Esselstyn CB Jr. Updating a 12-year experience with arrest and reversal therapy for coronary heart disease (an overdue requiem for palliative cardiology). Am J Cardiol. 1999 Aug 1;84(3):339-41, A8. doi: 10.1016/s0002-9149(99)00290-8. PMID 10496449
- [Background] Nicholson AS, Sklar M, Barnard ND, Gore S, Sullivan R, Browning S. Toward improved management of NIDDM: A randomized, controlled, pilot intervention using a lowfat, vegetarian diet. Prev Med. 1999 Aug;29(2):87-91. doi: 10.1006/pmed.1999.0529. PMID 10446033